CLINICAL TRIAL: NCT00089206
Title: Vaccination With Synthetic Melanoma Peptides Administered With GM-CSF-in-Adjuvant in Patients With Advanced Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Craig L Slingluff, Jr, Professor of Surgery, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10049; UVACC-MEL-42; UVACC-24802
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma; recurrent intraocular melanoma; iris melanoma; extraocular extension melanoma; ciliary body and choroid melanoma, medium/large size
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — incomplete Freund's adjuvant; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: incomplete Freund's adjuvant
Biological: multi-epitope melanoma peptide vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor immune response in patients with unresectable stage III or IV melanoma treated with vaccine comprising multiple synthetic melanoma peptides, sargramostim (GM-CSF), and Montanide ISA-51.

OUTLINE: Patients receive vaccine comprising multiple synthetic melanoma peptides, sargramostim (GM-CSF), and Montanide ISA-51 on days 1, 8, 15, 29, 36, and 43. Patients undergo removal of the lymph node draining the vaccination site on day 22 to assess immune response.

PROJECTED ACCRUAL: A maximum of 29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Unresectable stage III or IV disease
  * Mucosal or ocular disease allowed
* Positive HLA-A1, -A2, or -A3 expression

PATIENT CHARACTERISTICS:

Age

* 12 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL

Hepatic

* Liver function tests ≤ 2.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Weight ≥ 100 pounds
* Not pregnant or nursing
* No other malignancy within the past 5 years except squamous cell or basal cell skin cancer without known metastasis, carcinoma in situ of the breast, or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior vaccination with any of the peptides used in this protocol
* More than 1 year since prior melanoma vaccine therapy
* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior growth factors
* More than 4 weeks since prior allergy shots

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior steroid therapy

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Prior tumor resection allowed

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-08; Primary Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Study Chair — University of Virginia
Locations (1):
- Cancer Center at the University of Virginia, Charlottesville, Virginia, United States